CLINICAL TRIAL: NCT03497650
Title: Unilateral Strength Training and Mirror Therapy for Enhancing Lower Limb Motor Function Post Stroke: A Pilot Randomised Controlled Trial
Brief Title: Unilateral Strength Training and Mirror Therapy for Chronic Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Technology, Sligo (Other)
Responsible Party: Principal Investigator, Dr. John Bartlett, Head of Research, Institute of Technology, Sligo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ITSligo Daniel Simpson
Record Dates: First submitted 2018-03-24; First posted 2018-04-13 (Actual); Last update posted 2018-04-13 (Actual); Status verified 2018-04

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Mirror Movement Therapy

STUDY DESIGN:
Intervention Model Description: Pilot Randomised Controlled Trial
Who Masked: Outcomes Assessor
Masking Description: Outcome assessor only was masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mirror Therapy + Cross-Education. (Experimental): Patients performed 4 sets of 5 maximal isometric ankle dorsiflexions with their less-affected lower limb while observing the reflection of the exercising limb in the mirror which was placed in the patient's mid-sagittal plane. Training sessions took place 3 days per week for four weeks in the participant's own home under the supervision of 2 exercise professionals.
  Interventions: Device: Mirror Therapy; Other: Cross-Education of Strengthening.
- Cross-Education of Strengthening. (Active Comparator): Patients trained without a mirror entirely. They performed 4 sets of 5 maximal isometric ankle dorsiflexions with their less-affected lower limb. Training sessions took place 3 days per week for four weeks in the participant's own home under the supervision of 2 exercise professionals.
  Interventions: Other: Cross-Education of Strengthening.

INTERVENTIONS:
Device: Mirror Therapy — Mirror Therapy involved the patient sitting on a chair with a standard mirror placed between both legs with the reflective side of the mirror facing the non-affected leg. The patient is instructed to observe the reflection of the non-affected limb during the sessions. The patient was not given any instruction on the use of the affected limb.
  Arms: Mirror Therapy + Cross-Education.
Other: Cross-Education of Strengthening. — Cross-education of strengthening involves training one side of the body with the intention of producing strengthening gains on both sides of the body. In this case the strengthening was done on the non-affected leg of each stroke patient.

SUMMARY:
This is a pilot randomised controlled trial investigating a combination of unilateral strength training (cross-education) and mirror therapy for the rehabilitation of lower limb impairment following a stroke. This study has been conducted as part of a PhD qualification at the Institute of Technology Sligo in Ireland with all assessments being conducted at the institute and all therapy sessions taking place at the participant's home. The study was conducted in conjunction with Sligo University Hospital and it attained ethical approval through the relevant University Hospital Ethics Committee.

DETAILED DESCRIPTION:
The study necessitated patients with chronic stroke to perform a strength training programme with their less-affected lower limb. The mirror and strength training group observed the reflection of the training limb in a mirror, the strength training only group exercised without a mirror entirely. Patients were referred through Hospital Health Professionals. Prior to trial commencement all participants were given comprehensive trial information and provided signed written informed consent. A total of 35 participants were recruited. After a warm-up participants performed 4 sets of 5 maximal isometric ankle dorsiflexion contractions with their less-affected lower limb, three days per week, for four weeks. Patients received outcome assessment prior to the beginning of the intervention, directly after it and at three-month follow-up assessment. All assessments were carried out by a blinded Chartered Physiotherapist specialising in stroke rehabilitation. Patients were assessed using established outcome measures for lower limb isometric strength, motor function, muscle tone, and self-perceived participation.

ELIGIBILITY:
Inclusion Criteria:

Chronic stroke diagnosed by a physician at least 6 months prior to study begin Discharged from formal rehabilitation services (not receiving outpatient rehabilitation on more than a monthly basis, but may still be in receipt of occupational or language therapy).

Exclusion Criteria:

Impaired cognition (Mini mental state examination (MMSE) < 21) Cardiovascular, neurological or musculoskeletal impairments of the lower extremity not related to stroke that would prevent strength training.

Visual impairments that would interfere with the ability to participate safely in isometric training and observe mirror images.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2014-10-22 (Actual); Primary Completion 2017-08-16 (Actual); Study Completion 2017-08-16 (Actual)

PRIMARY OUTCOMES:
Maximal Isometric ankle dorsiflexion Strength. | 10 minutes
  Assessed with the Biodex System 3 Pro Isokinetic Dynamometer with the Biodex Advantage Software version 3.45 (Biodex Medical Systems, Inc., Shirley, New York, USA). Peak Torque, Rate of Torque Development and Average Torque over a single contraction was analysed. A higher torque measurement indicates a greater contraction strength.

SECONDARY OUTCOMES:
Modified Ashworth Scale (MAS). | 10 minutes.
  Muscle tone measure. Range 0 (No increase in muscle tone) to 4 (Affected part(s) rigid in flexion or extension).
Timed Up and Go (TUG). | 5 minutes.
  Assessment of the International Classification of Functioning, Disability and Health activity level. Used to measure basic mobility and balance manoeuvres; the ability to perform sequential motor tasks relative to walking and turning. Minimal Detectable Change = 2.9 seconds. A faster time indicates better functional ability.
10 Metre Walk Test (10MWT). | 5 minutes.
  Assessment of the International Classification of Functioning, Disability and Health activity level. Used to assess walking velocity in metres per second (m/s) over a short duration. Lower times indicate an increased walking velocity. Minimal Clinically Important Difference (MCID) is reported as; Small meaningful change = 0.06 m/s and Substantial meaningful change = 0.14 m/s. A higher score indicates a faster walking velocity.
London Handicap Scale (LHS). | 10 minutes
  Measurement of self-perceived impact of stroke over 6 domains of a patient's life (mobility, physical independence, occupation, social integration, orientation, and economic self - sufficiency). Scoring range of 0 to 1, where a score of 1 indicated 'No Disadvantage and a score of 0 indicates 'most severe disadvantage'.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Simpson, PhD, Principal Investigator — IT Sligo
Locations (1):
- Institute of Technology, Sligo, Sligo, Co Sligo, Ireland

IPD SHARING:
Plan to Share IPD: No
No IPD is shared with any other researchers.

DOCUMENTS (3):
  • Study Protocol (2015-07-12): https://cdn.clinicaltrials.gov/large-docs/50/NCT03497650/Prot_000.pdf
  • Statistical Analysis Plan (2015-07-12): https://cdn.clinicaltrials.gov/large-docs/50/NCT03497650/SAP_001.pdf
  • Informed Consent Form (2015-07-12): https://cdn.clinicaltrials.gov/large-docs/50/NCT03497650/ICF_002.pdf